CLINICAL TRIAL: NCT00476450
Title: Effects of Peripheral Blood Stem Cell Transplantation on the Microbial Flora of the Oral Cavity
Brief Title: Effects of Stem Cell Transplantation on Bacteria in the Mouth
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 070153; 07-CC-0153
Record Dates: First submitted 2007-05-19; First posted 2007-05-22 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-03-07

CONDITIONS: Allogeneic Peripheral Blood Stem Cell Transplant
Keywords: Oral Microbial Flora; Hematopoietic Stem Cell Transplant; Allogeneic Stem Cell Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
This study will examine bacteria in patients mouths at different times during stem cell transplantation and recovery. Drugs patients receive as part of the conditioning process for a stem cell transplant increase their risk of infection. There might be a link between the bacteria in the mouth and the bacteria that can cause infections. Knowing the changes in bacteria might help researchers determine the best method to prevent infections.

Patients 18 years of age and older who are scheduled to receive a stem cell transplant may be eligible for this study.

Participants undergo the following procedures:

Review of medical records

Interview about their oral care

Oral examination

Collection of oral specimens just before the stem cell transplant, immediately after the transplant, and 3 weeks after the transplant. The specimens are obtained as follows:

* <TAB>-About one-fourth teaspoon of saliva is collected with a suction device similar to that used in a dental office.
* <TAB>-Plaque from the surface of a tooth is collected with a plastic toothpick.
* <TAB>-Skin cells from the inside of the cheek and the surface of the tongue are collected with a small soft brush.
* <TAB>-If a tube is inserted into the patient s lungs to assist breathing and the patient is admitted to the intensive care unit, a specimen from the lungs is collected.

Patients are followed for 100 days after their transplant. Additional oral specimens are obtained from those who develop signs and symptoms of respiratory infection.

DETAILED DESCRIPTION:
The mouth is a complex biological ecosystem normally containing over 700 different species of bacteria. These bacteria live in an exopolysacchride matrix biofilm. Usually, bacteria colonize the oral cavity benignly. However, there are several studies in critically ill patients demonstrating changes in oral flora with acute illness. Identification of respiratory pathogens in the mouth has led researchers to hypothesize that a relationship exists between the oral cavity and pulmonary infections. A common complication of allogeneic peripheral blood stem cell transplant (PBSCT) is infection and pneumonia. Identification of potential pathogens in the oral cavity of allogeneic stem cell patients could indicate a similar association between oral pathogens and infection. A few studies describe the oral microbial community in these patients and the possibility that these organisms are a source of infection.

The primary objective of this study is to describe the changes in oral microbial flora of allogeneic SCT patients at three time points during their treatment and recovery. Observed differences in microbial organisms from baseline (prior to transplantation), through neutropenia (within 48 hours of nadir post-transplantation) and myeloid engraftment (14-21 days post transplantation) will be described.

In the course of their treatment, if patients develop respiratory signs and symptoms that require either a re-admission to an inpatient unit or intensive care unit admission, then additional oral specimens will be collected.

The secondary objective is to assess the oral microbial flora found after development of respiratory signs and symptoms in allogeneic PBSCT patients in the first 100 days post-transplant. In addition, if the patient requires intubation, tracheal aspirates and oral specimens will be collected.

The population is composed of adult patients who are planning to undergo an allogeneic PBSCT and can provide informed consent. The design is a prospective, descriptive study of the microbial flora of the oral cavity of adult allogeneic stem cell transplant patients. Saliva specimens, dental plaque and mucosal brushings will be collected at the three different times. Oral specimens will be obtained from patients who develop respiratory signs or symptoms that require an additional inpatient or intensive care unit admission. Patients will be followed and assessed for respiratory signs, symptoms, inpatient or ICU admission until day 100 post-transplant. The presence of bacteria (type and species) will be determined by molecular genetics. The identification of bacteria will be studied using various comparative molecular techniques, including DNA arrays and Real-Time Polymerase Chain Reaction (RT-PCR).

ELIGIBILITY:
* INCLUSION CRITERIA:

All adult patients admitted to the Clinical Research Center of the NIH who are 18 years of age or older who are scheduled to undergo an allogeneic PBSCT are eligible for enrollment. Collection of oral specimens in children who are allogeneic transplant recipients would increase the anxiety in these participants and may require sedation. For this reason children will be excluded from this protocol.

All adult patients who provide informed consent and who are scheduled to receive an allogeneic bone marrow transplant are eligible for enrollment.

EXCLUSION CRITERIA:

Patients who have had recent oral surgery or oral trauma will be excluded.

Patients with tracheostomies will also be excluded.

Patients with sickle cell disease or chronic granulomatous disease who are being transplanted will be excluded from the protocol.

Patients who are less than 18 years of age will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-05-16; Study Completion 2016-03-07

PRIMARY OUTCOMES:
Description of the oral microbiome | Baseline, nadir of ANC and engraftment.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ames, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Socransky SS, Haffajee AD. Periodontal microbial ecology. Periodontol 2000. 2005;38:135-87. doi: 10.1111/j.1600-0757.2005.00107.x. No abstract available. PMID 15853940
- [Background] Mager DL, Ximenez-Fyvie LA, Haffajee AD, Socransky SS. Distribution of selected bacterial species on intraoral surfaces. J Clin Periodontol. 2003 Jul;30(7):644-54. doi: 10.1034/j.1600-051x.2003.00376.x. PMID 12834503
- [Background] Kolenbrander PE, Andersen RN, Blehert DS, Egland PG, Foster JS, Palmer RJ Jr. Communication among oral bacteria. Microbiol Mol Biol Rev. 2002 Sep;66(3):486-505, table of contents. doi: 10.1128/MMBR.66.3.486-505.2002. PMID 12209001